CLINICAL TRIAL: NCT01353170
Title: Comparison Among Different Dialysate Calcium Concentrations in Bicarbonate Hemodialysis
Brief Title: Calcium Concentration in Bicarbonate Hemodialysis (HD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miulli General Hospital (Other)
Responsible Party: Carlo Basile M D, Miulli GH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Basile calcium
Record Dates: First submitted 2011-05-09; First posted 2011-05-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2010-12

CONDITIONS: Calcium Mass Balances and Serum Calcium Profiling in hd Patients
Keywords: Serum calcium; Dialysate; Mass balance; Blood pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prevalent hd patients (Experimental): Patients undergoing three consecutive cross-over hd session with 3 different dialysate calcium concentrations
  Interventions: Other: Dialysate calcium concentration

INTERVENTIONS:
Other: Dialysate calcium concentration — Calcium dialysate concentrations: 1.25, 1.35 and 1.5 mmol/l

SUMMARY:
The study was designed in order to investigate the effects of 3 different dialysate calcium concentrations may exert on mineral metabolism and hemodynamic stability in standard hemodialysis (hd).

ELIGIBILITY:
Inclusion Criteria:

* bicarbonate hd since 6 months
* uncomplicated hd sessions

Exclusion Criteria:

* Incident patients
* unstable hd patients
* patients aged less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Serum calcium concentrations | 4 hours
  Evaluation of calcium mass balances and ionized calcium serum concentrations profiling during three hd sessions with different calcium concentrations in the dialysate

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology and dialysis unit Miulli General Hospital, Acquaviva delle Fonti, Bari, Italy